CLINICAL TRIAL: NCT03069365
Title: A Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Glecaprevir/Pibrentasvir in Renally-Impaired Adults With Chronic Hepatitis C Virus Genotype 1 - 6 Infection (EXPEDITION-5)
Brief Title: A Study to Evaluate the Efficacy and Safety of Glecaprevir/Pibrentasvir in Adults With Chronic Hepatitis C Virus Genotype 1 - 6 Infection and Renal Impairment
Acronym: EXPEDITION-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-127; 2016-004182-60 (EudraCT Number)
Expanded Access: NCT03123965 (Approved for marketing)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Chronic Hepatitis C Virus; Chronic Kidney Disease; Glecaprevir; Pibrentasvir; Hepatitis C Virus Genotype; Compensated cirrhosis; Non-cirrhotic; Interferon (IFN); Treatment naïve; Sofosbuvir (SOF); Pegylated interferon (pegIFN); Ribavirin (RBV)
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Renal Insufficiency, Chronic | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- GLE/PIB for 8 weeks (Experimental): HCV genotype 1,2,4-6 non-cirrhotic, treatment-naive or treatment-experienced; genotype 3 non-cirrhotic, treatment-naïve participants treated with glecaprevir/pibrentasvir (GLE/PIB): three 100 mg/40 mg co-formulated tablets once daily with food for 8 weeks
  Interventions: Drug: Glecaprevir/pibrentasvir
- GLE/PIB for 12 weeks (Experimental): HCV genotype 1,2,4-6 compensated cirrhosis, treatment-naive or treatment-experienced; genotype 3 compensated cirrhosis, treatment- naïve participants treated with glecaprevir/pibrentasvir (GLE/PIB): three 100 mg/40 mg co-formulated tablets once daily with food for 12 weeks
  Interventions: Drug: Glecaprevir/pibrentasvir
- GLE/PIB for 16 weeks (Experimental): HCV genotype 3 non-cirrhotic or with compensated cirrhosis, treatment-experienced participants treated with glecaprevir/pibrentasvir (GLE/PIB): three 100 mg/40 mg co-formulated tablets once daily with food for 16 weeks
  Interventions: Drug: Glecaprevir/pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/pibrentasvir — Film-coated tablet
  Other Names: ABT-493/ABT-530; MAVYRET

SUMMARY:
This was a Phase 3b, open-label, non-randomized, multicenter study to evaluate the efficacy and safety of glecaprevir/pibrentasvir (GLE/PIB) in participants with chronic hepatitis C virus (HCV) genotype (GT) 1 - 6 infection without liver cirrhosis or with compensated liver cirrhosis and with chronic renal impairment in participants who were either HCV treatment-naïve (TN) or prior treatment-experienced (TE) with interferon (IFN) or pegylated interferon (PegIFN) with or without ribavirin (RBV), or sofosbuvir (SOF) plus RBV with or without pegIFN.

DETAILED DESCRIPTION:
The study included a 42-day screening period, a treatment period of either 8, 12, or 16 weeks, and a 24-week post-treatment period. The duration of treatment was determined by product labeling. Participants received glecaprevir/pibrentasvir (GLE/PIB) 300 mg/120 mg once daily. Participants who completed or prematurely discontinued the treatment period were followed for 24 weeks after their last dose of study drug to monitor safety, hepatitis C virus ribonucleic acid (HCV RNA), and the emergence and persistence of viral substitutions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (of non-childbearing potential or using allowed contraceptive methods) at least 18 years of age time of Screening
* Participant had a positive anti-hepatitis C virus (HCV) antibody (Ab) and plasma HCV ribonucleic acid (RNA) greater than or equal to 1000 IU/mL at the Screening Visit.
* Participant had an estimated glomerular filtration rate (eGFR) less than 45 mL/min/1.73 m^2 as estimated by the Modification of Diet in Renal Disease (MDRD) method at Screening according to the following formula: eGFR (mL/min/1.73 m^2 ) = 175 × (Serum Creatinine) ^-1.154 × Age^-0.203 × (0.742 if female) × (1.212 if black), or were dialysis dependent. Subjects requiring dialysis had to have been receiving dialysis for at least 1 month prior to enrollment, and may have been on hemodialysis or peritoneal dialysis.
* Cirrhotic participants only: absence of hepatocellular carcinoma (HCC) as indicated by a negative ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI) within 3 months prior to Screening or a negative ultrasound at Screening. Participants who had an ultrasound with results suspicious of HCC followed by a subsequent negative CT or MRI of the liver were eligible for the study.

Exclusion Criteria:

* Female participants who were pregnant, breastfeeding, or were considering becoming pregnant during the study or for approximately 30 days after the last dose of study drug
* Current hepatitis B virus (HBV) or human immunodeficiency virus (HIV) infection on screening tests, defined as:
* Positive test result at Screening for hepatitis B surface antigen (HBsAg), or;
* HBV deoxyribonucleic acid (DNA) greater than lower limit of quantification (LLOQ) in participants with isolated positive hepatitis B core antibody (HBcAb), (i.e., negative HBsAg and Anti-HBsAg), or;
* Positive anti-HIV antibody (Ab).
* Any current or historical clinical evidence of decompensated cirrhosis, including any current or past evidence of Child-Pugh B or C classification, hepatic encephalopathy or variceal bleeding; radiographic evidence of small ascites; or prior or current empiric use of lactulose/rifaximin for neurologic indications. Prophylactic use of beta blockers was not exclusionary.
* Clinical history of acute renal failure in the 3 months prior to Screening
* History of severe, life-threatening, or other significant sensitivity to any excipients of the study drugs
* Clinically significant abnormalities or co-morbidities, or recent (within 6 months prior to study drug administration) alcohol or drug abuse that could preclude adherence to the protocol in the opinion of the investigator
* Receipt of any investigational or commercially available direct acting anti-HCV agents other than sofosbuvir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (38):
- United States (11):
  - Scripps Clinic /ID# 159116, La Jolla, California
  - Huntington Medical Foundation /ID# 160653, Pasadena, California
  - Tampa General Medical Group /ID# 159115, Tampa, Florida
  - Northwest Louisiana Nephrology /ID# 160652, Shreveport, Louisiana
  - Massachusetts General Hospital /ID# 159114, Boston, Massachusetts
  - North Shore University Hospital /ID# 159108, New Hyde Park, New York
  - Columbia Univ Medical Center /ID# 159112, New York, New York
  - Carolinas Medical Center /ID# 159113, Charlotte, North Carolina
  - University of Pennsylvania /ID# 159117, Philadelphia, Pennsylvania
  - Thomas Jefferson University /ID# 159754, Philadelphia, Pennsylvania
  - TX Liver Inst, Americ Res Corp /ID# 159111, San Antonio, Texas
- Canada (4):
  - Zeidler Ledcor Centre /ID# 160600, Edmonton, Alberta
  - Vancouver ID Research and Care /ID# 160598, Vancouver, British Columbia
  - GIRI Gastrointestinal Research Institute /ID# 160599, Vancouver, British Columbia
  - Toronto General Hospital /ID# 160601, Toronto, Ontario
- Germany (4):
  - Universitatsklinikum Mannheim /ID# 160829, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Frankfurt /ID# 160826, Frankfurt am Main, Hesse
  - Med Hochschule Hanover /ID# 160827, Hanover
  - Univ Johannes Gutenberg /ID# 160828, Mainz
- Greece (4):
  - General Hospital of Athens Laiko /ID# 160725, Athens, Attica
  - Gen Univ Hosp Alexandroupolis /ID# 160724, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 160726, Athens
  - Bioclinic Thessaloniki /ID# 160723, Thessaloniki
- Italy (4):
  - A.O.U. Policlinico S.Orsola-Malpighi /ID# 163349, Bologna, Emilia-Romagna
  - Policlinico A. Gemelli /ID# 160719, Rome, Lazio
  - Policlinico Paolo Giaccone /Id# 160718, Palermo, Sicily
  - A.O. Uni Giovanni e Ruggi /ID# 160720, Salerno
- Poland (2):
  - HepID - Diagnostyka I Terapia /ID# 161083, Lublin, Lublin Voivodeship
  - Uniwersytecki Szpital Kliniczn /ID# 161081, Bialystok
- Puerto Rico (2):
  - VA Caribbean Healthcare System /ID# 160754, San Juan
  - School of Medicine University of Puerto Rico-Medical Sciences Campus /ID# 160755, San Juan
- South Korea (3):
  - Hanyang University Seoul Hospi /ID# 160259, Seongdong, Seoul Teugbyeolsi
  - Severance Hospital /ID# 160261, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 160260, Seoul
- Spain (3):
  - Hospital Regional de Malaga /ID# 159976, Málaga, Malaga
  - Hospital Parc de Salut del Mar /ID# 159975, Barcelona
  - Hospital Universitario Doce de /ID# 159974, Madrid
- Karolinska Uni /ID# 159523, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brown RS Jr, Collins MA, Strasser SI, Emmett A, Topp AS, Burroughs M, Ferreira R, Feld JJ. Efficacy and Safety of 8- or 12 Weeks of Glecaprevir/Pibrentasvir in Patients with Evidence of Portal Hypertension. Infect Dis Ther. 2022 Apr;11(2):913-924. doi: 10.1007/s40121-022-00599-8. Epub 2022 Feb 17. PMID 35174470
- [Derived] Lawitz E, Flisiak R, Abunimeh M, Sise ME, Park JY, Kaskas M, Bruchfeld A, Worns MA, Aglitti A, Zamor PJ, Xue Z, Schnell G, Jalundhwala YJ, Porcalla A, Mensa FJ, Persico M. Efficacy and safety of glecaprevir/pibrentasvir in renally impaired patients with chronic HCV infection. Liver Int. 2020 May;40(5):1032-1041. doi: 10.1111/liv.14320. Epub 2019 Dec 26. PMID 31821716

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent to treat population: all participants who received at least 1 dose of study drug
Groups:
- GLE/PIB for 8, 12, or 16 Weeks: Glecaprevir/pibrentasvir (GLE/PIB): three 100 mg/40 mg co-formulated tablets once daily with food
Period: Overall Study
Arm/Group | GLE/PIB for 8, 12, or 16 Weeks
Started | 101
Completed | 100
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population: all participants who received at least 1 dose of study drug
Arm/Group | GLE/PIB for 8, 12, or 16 Weeks
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.03 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 74
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks Post Dosing (SVR12)
Description: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (LLOQ) 12 weeks after the last actual dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent to treat population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were counted as non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GLE/PIB for 8, 12, or 16 Weeks
Number analyzed (Participants) | 101
percentage of participants | 97.0 [91.6 to 99.0]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as:
  * Confirmed increase from nadir in hepatitis C virus ribonucleic acid (HCV RNA) defined as confirmed increase of > 1 log (subscript)10(subscript) IU/mL above nadir during treatment; or
  * Confirmed HCV RNA greater than or equal to 100 IU/mL after HCV RNA less than the lower limit of quantification (LLOQ) during study drug treatment; or
  * HCV RNA ≥ LLOQ at the end of treatment with at least 6 weeks of treatment
Time Frame: Up to 16 weeks
Population: Intent to treat population: all participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GLE/PIB for 8, 12, or 16 Weeks
Number analyzed (Participants) | 101
percentage of participants | 0 [0.0 to 3.7]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed hepatitis C virus ribonucleic acid (HCV RNA) ≥ the lower limit of quantification (LLOQ) between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment as planned with HCV RNA < LLOQ at the end of treatment and had post-treatment HCV RNA data; participants who had been shown to be reinfected were not considered to have relapsed.
  .
Time Frame: Up to 12 weeks after the last dose of study drug
Population: Intent to treat population: all participants who received at least 1 dose of study drug and who completed treatment, had HCV RNA < LLOQ at final treatment visit, and had at least one post-treatment HCV RNA value
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GLE/PIB for 8, 12, or 16 Weeks
Number analyzed (Participants) | 98
percentage of participants | 0 [0.0 to 3.8]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 20 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | GLE/PIB for 8, 12, or 16 Weeks
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 12/101
Other Adverse Events (participants affected / at risk) | 27/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLE/PIB for 8, 12, or 16 Weeks (N=101)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MYELOPATHY (Nervous system disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
EXTREMITY NECROSIS (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 (1)
VENOUS STENOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLE/PIB for 8, 12, or 16 Weeks (N=101)
PRURITUS (Skin and subcutaneous tissue disorders) | 16 (16)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 6 (6)
HYPERTENSION (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03069365/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03069365/SAP_001.pdf